CLINICAL TRIAL: NCT01238107
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Phase II Clinical Study to Evaluate Doses of MT-102 in Subjects With Cachexia Related to Stage III and IV Non-small Cell Lung Cancer and Colorectal Cancer
Brief Title: A Clinical Study With MT-102 in Subjects With Cancer Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Collaborators: Veeda Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-102-2001
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Cancer Cachexia
Keywords: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose (Experimental)
  Interventions: Drug: MT-102
- Low dose (Experimental)
  Interventions: Drug: MT-102
- Placebo (Placebo Comparator)
  Interventions: Drug: MT-102

INTERVENTIONS:
Drug: MT-102 — BETA BLOCKER

SUMMARY:
A phase II clinical study to evaluate MT-102 administered over a sixteen week period in subjects with cachexia related to non-small cell lung cancer and colorectal cancer

DETAILED DESCRIPTION:
Cachexia is a wasting disease, associated with significant morbidity and mortality, accompanying a wide range of serious illnesses, for which there are currently no widely approved therapeutic agents. Cachexia is defined as weight loss, associated with a chronic underlying disease, of at least 5% in 12 months or less. It is associated with fatigue, loss of muscle strength, a low fat free index and neurohormonal and biochemical abnormalities.

Cancer cachexia occurs in about a third of all patients with cancer and has been estimated to be the direct cause of death in up to 20% of all cancer related deaths. As with other solid tumours, colorectal cancer (CRC) and non-small cell lung cancer (NSCLC) have relatively high incidences of cachexia, approximately 28% and 34% respectively.Through its combined pharmacological actions, MT-102 has a multi-functional effect upon three potential pharmacological targets, each of which is relevant for cancer cachexia

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients aged between 25 to 80 years of age and with a life expectancy of greater than 3 months as judged by the treating physician.

  2. Confirmed diagnosis of one of:

  a. Non-curative stage III or stage IV Colorectal Cancer (CRC) not suitable for surgery, or b. Non-curative stage III or stage IV Non-small Cell Lung Cancer (NSCLC) not suitable for surgery;

  3. Patients who are receiving or who have already received a course of chemotherapy, with or without radiotherapy or surgery, with one of the following regimes:

  a. For non-small cell lung cancer, a platinum based regimen b. For colorectal cancer, a 5FU or Irinotecan based regimen

  4. Cachexia with ongoing weight loss that in the opinion of the investigator is due to the underlying cancer.

  5. Evidence of cachexia as judged by one of:

  a. ≥5% documented weight loss in the previous 12 months; or b. A subjective report of weight loss in the previous 12 months and a recorded body mass index (BMI) less than 20.0 kg/m2 c. Ongoing documented weight loss of at least 1kg in the week prior to day 0; or 1.25kg in the 2 weeks prior to day 0, or 1.5kg in the 3 to 6 weeks prior to day 0; provided that BMI is not more than 25.

  6. At least two of the following:

  a. Subjective report of decreased muscle strength b. Subjective report of fatigue c. Subjective report of anorexia d. Abnormal biochemistry with one or more of the following: i. CRP > ULN (as per Central Lab normal value) ii. Anemia (< 12 g/dl) iii. Low serum albumin (< 3.2 g/dl) 7. Patients of childbearing potential must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives; an intrauterine device; male or female condoms; diaphragm or cervical cap with spermicide; or abstinence) prior to randomisation and must agree to continue using such precautions until the end of the 140 day safety follow up; 8. Willing and able to comply with the protocol and to complete the study period; 9. Willing to forego other forms of experimental treatment during the study; 10. Signed and dated informed consent, prior to receipt of any study medication or any study related procedures.

  11. ECOG performance status 0, 1 or 2 12. Able to complete the performance tests (SCP, SMWT, SPPB, HGS) at the screening visit and with two consecutive pre-randomisation SMWT results that differ by no more than 30% from each other 13. At least 80% compliant during the placebo run in period

Exclusion Criteria:

1. 1. Pregnancy or lactation at screen or baseline visit;
2. ≥20% weight loss in the previous 3 months or a BMI of less than 16 kg/m2
3. Age greater than 80 or less than 25 at baseline visit;
4. Scheduled to start any new course of chemotherapy or to undergo a change in present chemotherapeutic regimen during the dose escalation phase of the study (the first three weeks after randomisation);
5. Any surgical procedure within the past month or any planned surgical procedure;
6. Any mechanical obstruction of the alimentary canal;
7. Any history or evidence of intractable vomiting;
8. A history or clinical evidence of any hyperthyroidism, cirrhosis, hepatic failure, HIV, renal failure (as determined by a serum creatinine > 250µmol/l or > 2.83 mg/dl at screen) or active tuberculosis (as confirmed by sputum or other microbiological methods, within the last five years);
9. Any physical, medical, socioeconomic or other non-cancer related cause for simple starvation, muscle wasting or weight loss;
10. Receiving enteral tube feeding or parenteral nutrition at screening or baseline visit;
11. Any clinical evidence of ascites or significant oedema or significant pleural effusion at screening or baseline visit;
12. Current or planned treatment with

    1. Any oral adrenal corticosteroids (inhaled or topical steroids and short-term use of dexamethasone around the time of chemotherapy are acceptable);
    2. Beta adrenergic blockers,
    3. Non-dihydropyridine calcium antagonists (e.g. Verapamil, diltiazem),
    4. Alpha adrenergic blockers,
    5. Ivabradine (Coralan, Procoralan),
    6. 5HT agonists or antagonists e.g. SSRI's, , (short-term use around the time of chemotherapy are acceptable)
    7. MAOI's,
    8. Beta agonists, (short term or on-and -off use of inhaled broncho-dilators are acceptable)
    9. Amiodarone,
    10. Megestrol, Anabolic Steroids or any other prescription medication intended to increase appetite or to treat unintentional weight loss.
13. Treatment with any investigational drug therapy within 28 days prior to the screening visit;
14. Previous history of administration of pindolol or s-pindolol;
15. History of allergy or reaction to any component of the MT 102/study drug formulation;
16. History or presence of congestive heart failure (with LVEF <45%) or uncontrolled hypertension (with BP >160/95 mm Hg);
17. Use of a pacemaker, implantable defibrillator, or internalized metal stent;
18. Resting pulse rate less than 68 beats per minute or high degree conduction defect on the electrocardiogram;
19. A resting supine systolic blood pressure less than 100 mm Hg.
20. A history of bronchospasm and bronchial asthma;
21. History or diagnosis of brain metastases

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate the effect of a 10mg / bd dose of MT-102 in comparison to placebo on the rate of weight change over a sixteen week period in patients with cachexia related to underlying stage III and stage IV colorectal or non-small cell lung cancer | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kumar n Pradhash, MD, Principal Investigator — TATA MEMORIAL HOSPITAL , MUMBAI
Locations (18):
- Charite Hospital Virchow-Klinikum Campus, Berlin, State of Berlin, Germany
- India (9):
  - Kumaran Hospital Private Ltd, Kilpauk, Chennai
  - Dr Kamakshi Memorial Hospital, Pallikaranai, Chennai
  - Vedanta Institute of Medical Science, Ahmedabad, Gujarat
  - Shree Krishna Hopsital, Anand, Gujarat
  - Kailash Cancer Hospital & Research Centre, Goraj, Gujarat
  - TATA Memorial Hopsital, Mumbai, Maharashtra
  - Curie Manavta Cancer Centre, Nashik, Maharashtra
  - Shatabdi Super Speciality Hospital, Nashik, Maharashtra
  - Noble Hopsital, Pune, Pune
- Malaysia (8):
  - Hospital Sultahan Bahiyah, Alor Star, Kedha
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Hospital Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Universiti Malaya Medical, Jalan Baharu, Kuala Lumpur
  - Tuanku Ja'afar Hospital, Seremban, Negeri Sembilan
  - International Islamic University Malaysia, Kuantan, Pahang
  - Penang General Hopsital, Pulau Pinang, Pulau Pinang
  - Hospital Umum Sarawak, Kuching, Sarawak